CLINICAL TRIAL: NCT02725385
Title: Stress and Coping in Caregivers of Pediatric Cancer Patients
Brief Title: Stress and Coping in Caregivers of Younger Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00025224; NCI-2014-01878 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01413 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-02-22; First posted 2016-04-01 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Anxiety; Depression
Keywords: No Evidence of Disease
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (stress and coping): PART I:
  Participants complete a questionnaire that measures several psychological constructs including stress, anxiety, depression, coping mechanisms, uncertainty, positive and negative emotions, and life satisfaction over 15-30 minutes.
  PART II:
  Participants undergo a Trier Social Stress Test during a laboratory session over 1.5 hours.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Physiologic Testing; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Physiologic Testing — Undergo Trier Social Stress Test
  Other Names: Physiologic Test; Study of Physiologic Variables
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This research trial studies stress and coping in caregivers of younger patients with cancer. Learning how caregivers of children with cancer experience and cope with chronic stress may help to develop effective programs for reducing caregiver stress.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine how the experience of distress and use of positive emotion coping strategies by pediatric cancer caregivers differs from caregivers of children with no chronic illnesses.

II. To determine how relationships between positive coping strategies and caregiver distress change during the different phases of a child's illness.

III. To explore how chronic caregiver stress affects physiological reactivity to and recovery from an acute laboratory stressor.

IV. To explore how different positive coping mechanisms help chronically stressed caregivers recover from acute stressors and how these efficacies change during the different phases of the child's illness.

OUTLINE:

PART I:

Participants complete a questionnaire that measures several psychological constructs including stress, anxiety, depression, coping mechanisms, uncertainty, positive and negative emotions, and life satisfaction over 15-30 minutes.

PART II:

Participants undergo a Trier Social Stress Test during a laboratory session over 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak English
* Must serve as a primary caregiver of their child (ages 0-17) - as reported by the participant
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* (Part 1 and Part 2): Must not have a family member who has already participated in the study
* (Part 2): Must not be pregnant or have a history of cardiovascular disease, hypertension, pituitary disorder, or adrenal disorder
* CONTROL PARTICIPANTS: (Part 1 and Part 2): Participants must not have a child with a chronic illness (e.g., diabetes, asthma, multiple sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults serving as a primary caregiver of their child
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Level of Caregiver Distress as measured by multiple regressions analysis | Up to 1 year
  To examine whether coping styles alone predict psychosocial outcomes, a simple multiple regressions will be conducted with coping styles (approach and avoidant positive emotion coping strategies) as the predictors and the psychosocial outcomes as dependent variables. To examine whether treatment status moderates the impact of coping style on psychosocial outcomes, a multiple regressions with treatment status will be conducted, each coping style individually, and an interaction term of treatment status coping style in predicting each of the psychosocial outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Waugh, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina